CLINICAL TRIAL: NCT00771758
Title: A Randomized, Double-Blind, Placebo- and Oxycodone Immediate Release (IR)-Controlled Study of Tapentadol IR for the Treatment of Acute Pain Caused by Vertebral Compression Fractures Associated With Osteoporosis
Brief Title: Tapentadol IR vs Oxycodone IR vs Placebo in Acute Pain From Vertebral Compression Fracture Associated With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015064; KF5503/40
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Back Pain
Keywords: Vertebral compression fracture; Osteoporosis; Acute pain; Analgesic; Oxycodone; Tapentadol
MeSH Terms: conditions — Back Pain; Osteoporosis; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): tapentadol IR 50 or 75 mg capsule every 4 - 6 hr as needed for up to 10 days maximum daily dose 450 mg
  Interventions: Drug: tapentadol IR
- 002 (Experimental): oxycodone IR 5 or 10 mg capsule every 4 - 6 hr as needed for up to 10 days maximum daily dose 60 mg
  Interventions: Drug: oxycodone IR
- 003 (Placebo Comparator): placebo 1 capsule every 4 - 6 hr as needed for up to 10 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxycodone IR — maximum daily dose 450 mg
  Arms: 002
Drug: placebo — 5 or 10 mg capsule every 4 - 6 hr as needed for up to 10 days
  Arms: 003
Drug: tapentadol IR — 50 or 75 mg capsule every 4 - 6 hr as needed for up to 10 days
  Arms: 001

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of tapentadol immediate release (IR) as compared with placebo and oxycodone IR in patients with acute pain caused by vertebral compression fractures (VCF) associated with assumed osteoporosis for whom treatment with oral opioid analgesics is appropriate.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), multicenter, double-blind (neither the patient nor the physician know the study drug administered) study to determine the efficacy and safety of tapentadol immediate release (IR) as compared with placebo and oxycodone IR in approximately 625 patients with acute pain caused by vertebral compression fractures (VCFs) associated with assumed osteoporosis for whom treatment with oral opioid analgesics is appropriate. Patients will be randomized to receive multiple doses of tapentadol IR 50 or 75 milligrams (mg) or oxycodone IR 5 or 10 mg or placebo for up to 10 days. Screening/Randomization Visit (Visit 1): Potential patients with acute thoracolumbar pain with either new onset of pain or acute exacerbation of previous pain associated with a VCF will be identified. The acute pain episode must have started within 14 days of Visit 1. The study will be explained and informed consent will be obtained. Patients will either have had a radiographic procedure to confirm diagnosis of a VCF within 3 months prior to Visit 1 or will have a radiographic procedure (e.g., lateral vertebral x-ray or magnetic resonance imaging, etc) performed at Visit 1 as standard of care. Patients must have moderate to severe acute vertebral pain and must be appropriate candidates for pain management with an oral opioid analgesic. At Visit 1, patients must report both a qualifying average back pain intensity score in the last 24 hours related to the current episode and a qualifying current back pain intensity on an 11-point numerical rating scale (NRS) where 0=no pain and 10=pain as bad as you can imagine. Patients must also have a qualifying score on the Mini-Mental State Examination (MMSE) to be eligible for study participation. At Visit 1, patients will have laboratory assessments (including a urine drug screen), physical and back examinations and an electrocardiogram (ECG). Patients will also complete paper copies of the sleep quality, functionality and vomiting assessments (i.e., morning (AM) and evening (PM) Interactive Voice Response [IVR] system questions except satisfaction with treatment). In addition, patients will have physical performance assessed. Patients who have taken long-acting or controlled-release opioid therapy or immediate release CII opioid formulations (e.g., Opana IR, Percocet, Percodan, oxycodone IR, Dilaudid) within the 1 month prior to Visit 1 are not eligible for the study. Patients taking a CIII opioid formulation (e.g., Tylenol with Codeine) or any other analgesic medication (e.g., Non-steroidal anti-inflammatory drugs (NSAIDs) not previously described above will be eligible for study participation if they meet all study criteria (e.g., pain intensity score), unless they take the CIII > 5 days/week in the 1 month prior to Visit 1. After randomization all analgesic medications other than the study drug are prohibited except for NSAIDs taken for a condition other than chronic back pain, provided the patient has been taking a stable regimen for at least one month before screening and plans to continue throughout the study. Patients may take up to 2 pills (any form) of acetaminophen (e.g., Tylenol Extra-Strength) for pain other than back pain (e.g., headache, joint pain) once per day only. Subjects who take up to 325 mg/day aspirin for cardiovascular prevention will be permitted to enter the study provided they are on a stable dose for at least 1 month prior to study entry and plan to continue the same dose during the study. Double-Blind Treatment: Patients may be enrolled and randomized with laboratory and ECG results pending. If the results of any of these tests suggest the patient is not in good health, the patient will immediately be discontinued from the study. Patients meeting study entry criteria will be randomized in a double-blind fashion in a 2:2:1 ratio to receive tapentadol IR, oxycodone IR, or matching placebo every 4-6 hours during waking hours as needed for pain. The first dose of study drug will be one capsule of tapentadol IR 50 mg, oxycodone IR 5 mg or placebo. Most patients will take the first dose of study drug in the office at Visit 1. All patients will be instructed to call the IVR system to complete another assessment of current back pain intensity immediately before taking the first dose of study drug. This call will be made by the patient from the study site unless the first dose cannot be taken in the office, in which case the patient will make the call from home. Patients will be instructed to call the IVR system every morning and each evening to complete assessments related to back pain intensity and pain relief. Patients will also respond to IVR system questions related to sleep quality, patient satisfaction with treatment and functionality (AM only) and vomiting (PM only). Patients who discontinue prematurely for any reason will be instructed to contact the study site to complete final assessments, prior to taking supplemental pain medication if applicable, and to schedule a final study visit. During this call, site personnel will obtain current pain intensity and pain relief scores from the patient; these scores will be documented. Patients will begin treatment on Day 1 with one "lower dose" capsule of study drug (tapentadol IR 50 mg, oxycodone IR 5 mg, or matching placebo). For subsequent doses, patients may remain at the "lower dose" capsule (tapentadol IR 50 mg, oxycodone IR 5 mg, or matching placebo) or may choose to take the "higher dose" (tapentadol IR 75 mg, oxycodone IR 10 mg, or matching placebo) every 4 to 6 hours during waking hours as needed depending on their level of pain and tolerability of the study drug. The duration of treatment with study drug will be up to 10 days. Tapentadol IR 450 mg or oxycodone IR 60 mg is the maximum daily dose allowed. Patients who require supplemental medication for insufficient analgesia will be discontinued from the study and will be treated at the investigator's discretion. All patients will receive a telephone call from the study staff on Day 3. During this telephone call, site personnel will inquire about the patient's overall status. Patients will return to the study site on Day 10/End of Study for the final visit (Visit 2). Patients who have not discontinued from the study prior to the final visit will complete a final assessment of current pain intensity and pain relief (on paper). In addition, all patients will have physical functionality assessed. Patients and investigators will each complete a global assessment of study drug. The investigator will also respond to two ease-of-care questions. Vital signs will be obtained, safety assessments will be completed and study drug will be collected. All patients will have their post-study analgesia prescribed at the investigator's discretion. Tapentadol IR 50 or 75 mg, oxycodone IR 5 or 10 mg, or placebo for up to 10 days. The dose is every 4-6 hours, as needed for pain. Maximum dosage is 450 mg tapentadol or 60 mg oxycodone per day.

ELIGIBILITY:
Inclusion Criteria:

* Female (non-pregnant, non-lactating) and male
* new onset of pain or acute exacerbation of previous pain associated with a VCF within 14 days prior to Visit 1
* Radiographic confirmation of a VCF within 3 months prior to Visit 1 or a radiographic procedure performed at Visit 1
* Average back pain intensity score in the last 24 hours related to the current episode and a qualifying current back pain intensity score
* Qualifying score on the Mini-Mental Status Exam
* Able to verbalize and differentiate with regard to location and intensity of pain
* Medically stable
* Sexually active women must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control at study entry and throughout the trial
* Women of childbearing potential must have a negative urine pregnancy test at Visit 1
* Physically and mentally willing and able to adhere to the protocol requirements and its prohibitions and restrictions
* Sign an informed consent document

Exclusion Criteria:

* Neurological symptoms or deficits, or radiculopathy related to the VCF
* Taken any of the following in the month before Visit 1: long-acting or controlled-release opioid, immediate release Class II opioid formulations or Class III opioid formulation (e.g., Tylenol with Codeine) > 5 days/week
* Systemic steroid therapy within 3 months before Visit 1
* Anticonvulsants, monoamine oxidase inhibitors, tricyclic antidepressants, neuroleptics, or serotonin norepinephrine reuptake inhibitor within 2 weeks before randomization
* Major trauma to or infection in the fractured vertebrae in the 6 months preceding study
* Pain due to herniated nucleus pulposus, high energy trauma, severe spinal stenosis, bone tumor at the level(s) of pathology or known canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression with an ongoing pain level of >= 5
* Severe cardiopulmonary deficiencies
* Active systemic or local infection
* History of alcohol or drug abuse in the investigator's judgment based on medical history and physical examination
* Malignancy within the past 2 years, with the exception of basal cell carcinoma
* Concomitant autoimmune inflammatory conditions
* History of laboratory values reflecting severe renal insufficiency
* History of moderately or severely impaired hepatic function or alanine aminotransaminase or aspartate aminotransferase greater than 3 times the upper limit of normal.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (37):
- United States (37):
  - Haleyville, Alabama
  - Tallassee, Alabama
  - Peoria, Arizona
  - Tucson, Arizona
  - Encinitas, California
  - Los Gatos, California
  - Mission Viejo, California
  - Oakland, California
  - Roseville, California
  - San Diego, California
  - Studio City, California
  - Vista, California
  - Bradenton, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Miami Springs, Florida
  - Ormond Beach, Florida
  - Saint Cloud, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Peachtree, Georgia
  - Savannah, Georgia
  - Valdosta, Georgia
  - Bloomington, Illinois
  - South Bend, Indiana
  - Covington, Louisiana
  - Minneapolis, Minnesota
  - North Massapequa, New York
  - Hickory, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Marion, Ohio
  - Eugene, Oregon
  - Aiken, South Carolina
  - Houston, Texas
  - Mesquite, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this outpatient, multicenter study occurred between August 28, 2008 and December 9, 2009.
  The study was terminated prematurely due to slow enrollment after 108 of 600 subjects enrolled. Valid statistical conclusions cannot be made due to the low number of subjects.
Pre-assignment Details: The study consisted of a screening/randomization period (one day) and a double blind active treatment period (10 days).
Groups:
- Tapentadol IR: 50 or 75 mg capsule every 4 - 6 hr as needed for up to 10 days; maximum daily dose 450 mg.
- Oxycodone IR: 5 or 10 mg capsule every 4 - 6 hr as needed for up to 10 days; maximum daily dose 60 mg.
- Placebo: 1 capsule every 4 - 6 hr as needed for up to 10 days
Period: Overall Study
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Started | 44 | 43 | 21
Completed | 36 | 31 | 19
Not Completed | 8 | 12 | 2
Not completed — Adverse Event | 2 | 8 | 1
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 21 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 7 | 33
  >=65 years | 29 | 32 | 14 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (12.28) | 69.3 (13.26) | 69.6 (12.36) | 69.5 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 14 | 76
  Male | 14 | 11 | 7 | 32
Region of Enrollment [Number; unit: participants]
  USA | 44 | 43 | 21 | 108

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference Over 3 Days (SPID72)
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID72 was calculated as the time-weighted Sum of PID scores over 72 hours. The range of SPID72 is from -720 to 720. The higher value in SPID indicates greater pain relief.
  The study was terminated prematurely due to slow enrollment after 108 of 600 subjects enrolled. Valid statistical conclusions cannot be made due to the low number of subjects.
Time Frame: 3 Days (72 hours)
Population: The modified Intent-to-Treat(mITT) population was defined as all randomized patients who took at least one dose of study drug and had a baseline pain intensity assessment via the Interactive Voice Response (IVR) system with score ≥5 on an 11-point NRS.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 139.0 (132.57) | 129.4 (115.76) | 114.2 (99.87)

2. Secondary Outcome: 30% Responder Rate on Day 3.
Description: The 30% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 30% from baseline in pain intensity at Day 3 (average of Day 3 PM and Day 4 AM).
Time Frame: Day 3
Population: modified Intent-to-Treat (mITT) population defined as all randomized participants who took at least one dose of study drug and had a baseline pain intensity assessment via the Interactive Voice Response (IVR) system with score ≥5 on an 11-point NRS.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 36.1 | 39.0 | 50.0

3. Secondary Outcome: 50% Responder Rate on Day 3.
Description: The 50% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 50% from baseline in pain intensity at Day 3 (average of Day 3 PM and Day 4 AM).
Time Frame: Day 3
Population: modified Intent-to-Treat (mITT) population defined as all randomized participants who took at least one dose of study drug and had a baseline pain intensity assessment via the IVR system with score ≥5 on an 11-point NRS.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 25.0 | 24.4 | 25.0

4. Secondary Outcome: 30% Responder Rate on Day 5.
Description: The 30% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 30% from baseline in pain intensity at Day 5 (average of Day 5 PM and Day 6 AM).
Time Frame: Day 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 44.4 | 48.8 | 35.0

5. Secondary Outcome: 50% Responder Rate on Day 5.
Description: The 50% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 50% from baseline in pain intensity at Day 5 (average of Day 5 PM and Day 6 AM).
Time Frame: Day 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 25.0 | 26.8 | 25.0

6. Secondary Outcome: 30% Responder Rate on Day 10.
Description: The 30% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 30% from baseline in pain intensity at Day 10 (average of Day 9 PM and Day 10 AM).
Time Frame: Day 10
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 52.8 | 39.0 | 55.0

7. Secondary Outcome: 50% Responder Rate on Day 10.
Description: The 50% responder rate was defined as the proportion of participants with a value of percentage change greater than or equal to the 50% from baseline in pain intensity at Day 10 (average of Day 9 PM and Day 10 AM).
Time Frame: Day 10
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
percentage of participants | 30.6 | 26.8 | 30.0

8. Secondary Outcome: Sum of Pain Intensity Difference Over 2 Days (SPID48)
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID48 was calculated as the time-weighted Sum of PID scores over 48 hours. The range of SPID48 is from -480 to 480. The higher value in SPID indicates greater pain relief.
Time Frame: 2 Days (48 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 82.1 (92.13) | 86.5 (69.46) | 67.1 (66.66)

9. Secondary Outcome: Sum of Pain Intensity Difference Over 5 Days (SPID120)
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID120 was calculated as the time-weighted Sum of PID scores over 120 hours. The range of SPID120 is from -1200 to 1200. The higher value in SPID indicates greater pain relief.
Time Frame: 5 Days (120 hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 252.7 (208.91) | 227.1 (200.66) | 198.4 (177.76)

10. Secondary Outcome: Sum of Pain Intensity Difference Over 10 Days
Description: Pain Intensity (PI) was assessed on 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Pain Intensity Difference (PID) was the difference between baseline PI (prior to the first dose) and current PI at assessment. Sum of Pain Intensity Difference Over 10 Days was calculated as the time-weighted Sum of PID scores up to Day 10, 8 AM. The range is from -2160 to 2160. The higher value in Sum of Pain Intensity Difference indicates greater pain relief.
Time Frame: 10 Days (216 Hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 505.0 (373.00) | 422.9 (382.78) | 389.9 (343.31)

11. Secondary Outcome: Total Pain Relief (TOTPAR) Over 2 Days
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to hour 48. The range of TOTPAR over 2 days is from 0 to 192. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 2 Days (48 Hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 84.7 (38.79) | 92.3 (42.42) | 89.5 (44.55)

12. Secondary Outcome: Total Pain Relief (TOTPAR) Over 3 Days
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to hour 72. The range of TOTPAR over 3 days is from 0 to 288. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 3 Days (72 Hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 126.5 (57.98) | 138.3 (61.02) | 125.8 (66.12)

13. Secondary Outcome: Total Pain Relief (TOTPAR) Over 5 Days
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to hour 120. The range of TOTPAR over 5 days is from 0 to 480. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 5 Days (120 Hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 216.8 (97.36) | 232.6 (102.87) | 220.7 (106.00)

14. Secondary Outcome: Total Pain Relief (TOTPAR) Over 10 Days
Description: Pain Relief was defined as a 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum over all pain relief up to Day 10, 8 AM. The range of TOTPAR over 10 days is from 0 to 864. A higher value in TOTPAR indicated greater pain relief.
Time Frame: 10 Days (216 Hours)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 378.8 (167.27) | 414.4 (190.38) | 391.7 (184.35)

15. Secondary Outcome: Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) Over 2 Days
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 2 days is from -480 to 672. A higher value in SPRID indicated greater pain relief.
Time Frame: 2 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 168.6 (109.56) | 178.9 (97.04) | 158.9 (87.52)

16. Secondary Outcome: Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) Over 3 Days
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 3 days is from -720 to 1008. A higher value in SPRID indicated greater pain relief.
Time Frame: 3 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 265.5 (162.13) | 267.7 (152.74) | 240.0 (130.29)

17. Secondary Outcome: Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) Over 5 Days
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 5 days is from -1200 to 1680. A higher value in SPRID indicated greater pain relief.
Time Frame: 5 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 469.5 (270.72) | 459.7 (266.29) | 419.1 (229.41)

18. Secondary Outcome: Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) Over 10 Days
Description: The Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID) was derived from Sum of TOTPAR and SPID. The range of SPRID over 10 days is from -2160 to 3024. A higher value in SPRID indicated greater pain relief.
Time Frame: 10 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 36 | 41 | 20
Scores on a scale | 883.8 (482.19) | 837.3 (509.07) | 781.7 (442.17)

19. Secondary Outcome: Change From Baseline in Physical Performance: Measured Walk - Change in Distance Walked in the End of Study
Description: The participants were assessed whether were able to walk for 4 meters at each visit. For those subjects who were unable to walk 4 meters, the distance walked would be recorded. For those completed the walk, 4 meters were recorded. The change in distance walked at the end of study was derived using the distance walked at baseline minus the distance walked at the end of study (Day 10). The range of change in distance walked is from -4 to 4. A negative value indicated better performance.
Time Frame: Day 10
Population: Intent-to-Treat subjects.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
meters | -0.1 (0.32) | 0.4 (2.31) | 0.0 (0.00)

20. Secondary Outcome: Change From Baseline in Physical Performance: Measured Walk - Change in Time Taken Per Meter to Take Walk in the End of Study
Description: The time for the subject to walk for 4 meters was measured at baseline and the end of study. Change = baseline - end of study. For the change in each treatment group, only subjects who were assessed at both baseline and end of study were summarized. A positive value of Change indicated performance improved.
Time Frame: Day 10
Population: Intent-to-Treat subjects.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
seconds | 0.6 (2.10) | 3.5 (18.24) | 0.6 (1.72)

21. Secondary Outcome: Change From Baseline in Physical Performance: Chair Stand - Change in Number of Chair Stands Completed in the End of Study
Description: The participants were assessed whether were able to rise from a chair 5 times at each visit. For those subjects who were unable to complete all 5 rises, the number of rises would be recorded. For those completed the 5 rises, 5 were recorded. The change in number of chair stands at the end of study was derived using the number of chair stands at baseline minus the number of chair stands at the end of study (Day 10). The range of change in number of chair stands is from -5 to 5. A negative value indicated better performance.
Time Frame: Day 10
Population: Intent-to-Treat subjects.
Measure: Mean (Standard Deviation); unit: chair stands
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
chair stands | -0.1 (0.23) | -0.0 (0.16) | 0.0 (0.00)

22. Secondary Outcome: Change From Baseline in Physical Performance: Chair Stand - Change in Time Taken to Complete Chair Stands in the End of Study
Description: The time for the subject to rise from a chair 5 times was measured at baseline and the end of study.
  Change = baseline - end of study. For the change in each treatment group, only subjects who were assessed at both baseline and end of study were summarized. A positive value of Change indicated performance improved.
Time Frame: Day 10
Population: Intent-to-Treat subjects.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
second | 3.1 (9.51) | 3.6 (11.08) | 2.6 (9.22)

23. Secondary Outcome: Summary of Subject Satisfaction With Treatment on Day 2
Description: Treatment satisfaction was measured using a 7-point scale where 1 = very satisfied and 7 = very dissatisfied.
Time Frame: Day 2
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
Scores on a scale | 3.5 (1.58) | 3.0 (1.69) | 3.6 (2.23)

24. Secondary Outcome: Summary of Subject Satisfaction With Treatment on Day 3
Description: Treatment satisfaction was measured using a 7-point scale where 1 = very satisfied and 7 = very dissatisfied.
Time Frame: Day 3
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
Scores on a scale | 3.3 (1.69) | 2.8 (1.71) | 3.3 (1.70)

25. Secondary Outcome: Summary of Subject Satisfaction With Treatment on Day 5
Description: Treatment satisfaction was measured using a 7-point scale where 1 = very satisfied and 7 = very dissatisfied.
Time Frame: Day 5
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
Scores on a scale | 3.5 (1.72) | 2.6 (1.27) | 3.7 (1.60)

26. Secondary Outcome: Summary of Subject Satisfaction With Treatment on Day 10
Description: Treatment satisfaction was measured using a 7-point scale where 1 = very satisfied and 7 = very dissatisfied.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
Scores on a scale | 3.3 (1.94) | 2.5 (1.38) | 3.1 (1.61)

27. Secondary Outcome: Sleep Quality - Shift From Baseline to End of Study (Tapentadol IR)
Description: Sleep Quality was assessed by a 4-point numeric scale (1=excellent, 2=good, 3=fair, and 4=poor). The sleep question was "Please rate the overall quality of your sleep last night.", which was administered via Interactive Voice Response (IVR) system in the morning.
Time Frame: 10 days
Population: Tapentadol IR arm of Intent-to-Treat population. Shift table from baseline to end of study. Percentages were based on the number of intent-to-treat subjects within a screening category.
Measure: Number; unit: participants
Groups:
- Excellent - End of Study; Good - End of Study; Fair - End of Study; Poor - End of Study; Missing - End of Study; Baseline Total: Tapentadol IR
Arm/Group | Excellent - End of Study | Good - End of Study | Fair - End of Study | Poor - End of Study | Missing - End of Study | Baseline Total
Number analyzed (Participants) | 12 | 12 | 13 | 2 | 2 | 41
participants
  Excellent - Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Good - Baseline | 5 | 4 | 2 | 0 | 1 | 12
  Fair - Baseline | 2 | 8 | 8 | 1 | 0 | 19
  Poor - Baseline | 5 | 0 | 3 | 1 | 1 | 10
  Missing - Baseline | 0 | 0 | 0 | 0 | 0 | 0
  End of Study Total | 12 | 12 | 13 | 2 | 2 | 41

28. Secondary Outcome: Sleep Quality - Shift From Baseline to End of Study (Oxycodone IR)
Description: Sleep Quality was assessed by a 4-point numeric scale (1=excellent, 2=good, 3=fair, and 4=poor). The sleep question was "Please rate the overall quality of your sleep last night.", which was administered via IVR system in the morning.
Time Frame: 10 days
Population: Oxycodone IR arm of Intent-to-Treat population. Shift table from baseline to end of study. Percentages were based on the number of intent-to-treat subjects within a screening category.
Measure: Number; unit: participants
Groups:
- Excellent - End of Study; Good - End of Study; Fair - End of Study; Poor - End of Study; Missing - End of Study; Baseline Total: Oxycodone IR
Arm/Group | Excellent - End of Study | Good - End of Study | Fair - End of Study | Poor - End of Study | Missing - End of Study | Baseline Total
Number analyzed (Participants) | 9 | 13 | 12 | 6 | 3 | 43
participants
  Excellent - Baseline | 0 | 0 | 0 | 0 | 0 | 0
  Good - Baseline | 1 | 6 | 2 | 0 | 1 | 10
  Fair - Baseline | 8 | 6 | 7 | 3 | 0 | 24
  Poor - Baseline | 0 | 1 | 3 | 3 | 1 | 8
  Missing - Baseline | 0 | 0 | 0 | 0 | 1 | 1
  End of Study Total | 9 | 13 | 12 | 6 | 3 | 43

29. Secondary Outcome: Sleep Quality - Shift From Baseline to End of Study (Placebo)
Description: as for outcome 28
Time Frame: 10 days
Population: Placebo arm of Intent-to-Treat population. Shift table from baseline to end of study. Percentages were based on the number of intent-to-treat subjects within a screening category.
Measure: Number; unit: participants
Groups:
- Excellent - End of Study; Good - End of Study; Fair - End of Study; Poor - End of Study; Baseline Total: Placebo
Arm/Group | Excellent - End of Study | Good - End of Study | Fair - End of Study | Poor - End of Study | Baseline Total
Number analyzed (Participants) | 4 | 4 | 11 | 2 | 21
participants
  Excellent - Baseline | 0 | 0 | 0 | 0 | 0
  Good - Baseline | 2 | 0 | 3 | 0 | 5
  Fair - Baseline | 1 | 2 | 6 | 0 | 9
  Poor - Baseline | 1 | 2 | 2 | 2 | 7
  Missing - Baseline | 0 | 0 | 0 | 0 | 0
  End of Study Total | 4 | 4 | 11 | 2 | 21

30. Secondary Outcome: Summary of Functionality: Dressing - Proportion With at Least 2 Points of Improvement From Baseline to Day 2
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 2
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 14.7 | 8.6 | 11.1

31. Secondary Outcome: Summary of Functionality: Dressing - Proportion With at Least 2 Points of Improvement From Baseline to Day 3
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 3
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 19.4 | 13.9 | 15.8

32. Secondary Outcome: Summary of Functionality: Dressing - Proportion With at Least 2 Points of Improvement From Baseline to Day 5
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 5
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 25.0 | 14.8 | 11.1

33. Secondary Outcome: Summary of Functionality: Dressing - Proportion With at Least 2 Points of Improvement From Baseline to Day 10
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 28.6 | 25.0 | 7.1

34. Secondary Outcome: Summary of Functionality: Bath/Shower - Proportion With at Least 2 Points of Improvement From Baseline to Day 2
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 2
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 11.8 | 14.3 | 11.1

35. Secondary Outcome: Summary of Functionality: Bath/Shower - Proportion With at Least 2 Points of Improvement From Baseline to Day 3
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 3
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 16.7 | 19.4 | 10.5

36. Secondary Outcome: Summary of Functionality: Bath/Shower - Proportion With at Least 2 Points of Improvement From Baseline to Day 5
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 5
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 15.6 | 14.8 | 5.9

37. Secondary Outcome: Summary of Functionality: Bath/Shower - Proportion With at Least 2 Points of Improvement From Baseline to Day 10
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 21.4 | 20.8 | 7.1

38. Secondary Outcome: Summary of Functionality: Chair - Proportion With at Least 2 Points of Improvement From Baseline to Day 2
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 2
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 20.6 | 14.3 | 0

39. Secondary Outcome: Summary of Functionality: Chair - Proportion With at Least 2 Point of Improvement From Baseline to Day 3
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 3
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 16.7 | 8.3 | 10.5

40. Secondary Outcome: Summary of Functionality: Chair - Proportion With at Least 2 Points of Improvement From Baseline to Day 5
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 5
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 18.8 | 7.4 | 5.6

41. Secondary Outcome: Summary of Functionality: Chair - Proportion With at Least 2 Points of Improvement From Baseline to Day 10
Description: Level of functionality assessed using a 5-point scale where 0=no difficulty and 4=impossible without help.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percentage of participants | 28.6 | 8.3 | 14.3

42. Secondary Outcome: Patient Global Impression of Change (PGIC) at End of Study
Description: Patient Global Impression of Change (PGIC) was defined as the 7-point numeric scale, where 1=very much improved to 7=very much worse.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Number; unit: percenatage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percenatage of participants
  Very much improved | 17.1 | 9.3 | 9.5
  Much improved | 24.4 | 34.9 | 23.8
  Minimally improved | 26.8 | 34.9 | 23.8
  No change | 26.8 | 11.6 | 28.6
  Minimally worse | 0 | 4.7 | 4.8
  Much worse | 0 | 2.3 | 0
  Very much worse | 0 | 0 | 4.8

43. Secondary Outcome: Clinician Global Impression of Change (CGIC) at End of Study
Description: Clinician Global Impression of Change (CGIC) was defined as the 7-point numeric scale, where 1=very much improved to 7=very much worse.
Time Frame: Day 10
Population: Intent-to-Treat population.
Measure: Number; unit: percenatage of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percenatage of participants
  Very much improved | 19.5 | 7.0 | 14.3
  Much improved | 29.3 | 39.5 | 23.8
  Minimally improved | 19.5 | 34.9 | 33.3
  No change | 26.8 | 9.3 | 19.0
  Minimally worse | 0 | 4.7 | 4.8
  Much worse | 0 | 2.3 | 0
  Very much worse | 0 | 0 | 4.8

44. Secondary Outcome: Summary of Clinician Ease-of-Care at the End of Study: Time Comsuming
Description: The Clinician Ease-of-Care was defined on a 6-point scale, where 0 = "not at all" to 5="a very great deal."
Time Frame: Day 10
Population: Intent-to Treat population.
Measure: Number; unit: percent of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percent of participants
  Not at all | 51.2 | 51.2 | 47.6
  A little bit | 19.5 | 16.3 | 23.8
  Somewhat | 12.2 | 16.3 | 19.0
  Quite a bit | 12.2 | 9.3 | 4.8
  A great deal | 2.4 | 4.7 | 4.8
  A very great deal | 0 | 0 | 0

45. Secondary Outcome: Summary of Clinician Ease-of-Care at the End of Study: Bothersome
Description: The Clinician Ease-of-Care was defined on a 6-point scale, where 0 = "not at all" to 5="a very great deal."
Time Frame: Day 10
Population: Intent-to Treat population.
Measure: Number; unit: percent of participants
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Number analyzed (Participants) | 41 | 43 | 21
percent of participants
  Not at all | 56.1 | 53.5 | 76.2
  A little bit | 17.1 | 18.6 | 9.5
  Somewhat | 14.6 | 9.3 | 4.8
  Quite a bit | 7.3 | 14.0 | 4.8
  A great deal | 2.4 | 2.3 | 4.8
  A very great deal | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Tapentadol IR | Oxycodone IR | Placebo
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/43 | 0/21
Other Adverse Events (participants affected / at risk) | 23/44 | 29/43 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR (N=44) | Oxycodone IR (N=43) | Placebo (N=21)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol IR (N=44) | Oxycodone IR (N=43) | Placebo (N=21)
Nausea (Gastrointestinal disorders) | 15 | 19 | 1
Vomiting (Gastrointestinal disorders) | 12 | 19 | 4
Constipation (Gastrointestinal disorders) | 1 | 3 | 1
Dizziness (Nervous system disorders) | 8 | 7 | 0
Headache (Nervous system disorders) | 4 | 2 | 0
Somnolence (Nervous system disorders) | 4 | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0

LIMITATIONS AND CAVEATS:
Insufficient number of participants enrolled to meet proposed sample size, so that statistical inferences could not be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days